CLINICAL TRIAL: NCT06731374
Title: A Phase IV, Experimental Human Pneumococcal Challenge (EHPC) Model to Investigate Streptococcus Pneumoniae Serotype 3 (SPN3) Colonisation Following PCV15, a Double Blind Randomised Controlled Trial (DBRCT) in Healthy Participants Aged 18 - 50 Years in the UK.
Brief Title: Carriage to Assess Protection of New Pneumococcal Vaccines - PCV15
Acronym: RATIONALE-15
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Liverpool School of Tropical Medicine, United Kingdom (Unknown); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OVG 2024/02; MISP 101865 (Other Grant/Funding Number: Merck Sharp & Dohme (UK) Limited)
Record Dates: First submitted 2024-12-02; First posted 2024-12-12 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-11

CONDITIONS: Pneumococcal Disease; Pneumococcal Carriage
Keywords: Streptococcus pneumoniae; Experimental Human Pneumococcal Challenge; Pneumococcal carriage; PCV15; VAXNEUVANCE; SPN3
MeSH Terms: conditions — Pneumococcal Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCV-15 Vaccination (Experimental): One dose (0.5 ml) of PCV-15 is to be given Intramuscularly (IM) into the deltoid region of the arm at day 0.
  Interventions: Biological: PCV15; Biological: Streptococcus pneumoniae serotype 3
- Placebo (Placebo Comparator): 0.9% saline is to be given Intramuscularly (IM) into the deltoid region of the arm at day 0.
  Interventions: Biological: Streptococcus pneumoniae serotype 3; Biological: Placebo

INTERVENTIONS:
Biological: PCV15 — VAXNEUVANCE (Merck, Sharp & Dohme LLC, a subsidiary of Merck & Co, Inc., Rahway, NJ, USA [MSD]) is a 15-valent PCV containing capsular polysaccharides from serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 22F, and 33F adjuvanted with aluminium phosphate.
  Other Names: VAXNEUVANCE
  Arms: PCV-15 Vaccination
Biological: Streptococcus pneumoniae serotype 3 — Streptococcus pneumoniae SPN3 (Clade Ia, strain LIV014-S3) - Single inoculation at 80,000 colony-forming unit (CFU)/naris, 28 days after vaccination.
  Other Names: SPN3; pneumococcus serotype 3
Biological: Placebo — The placebo consists of 0.9% sodium chloride for injection
  Other Names: Saline Placebo; 0.9% Sodium Chloride
  Arms: Placebo

SUMMARY:
Streptococcus pneumoniae (pneumococcus) is a bacterium that causes just under four million serious infections every year. It is normal for pneumococcus bacteria to live in the noses of healthy adults and children as part of the nasal microflora without causing harm. This is called "carriage". But the bacteria can still be passed on to other people. If they are at-risk, for example elderly, or very young, or have pre-existing health conditions, the pneumococcus bacteria can cause pneumonia, which can cause serious life-threatening illness.

Pneumococcus bacteria are surrounded by a sugar capsule. But the capsule does not always have the same components. As a result, the bacteria are classified into more than 100 different types. To make them effective, the vaccines that are currently available contain the sugar capsules of the most common pneumococcal types that cause disease.

One such vaccine - PCV13 - has been effective globally in protecting against pneumococcus disease. It works because it controls the "carriage" (how a person carries the bacteria in their nose) of 13 types of the bacteria. Vaccines giving protection against other types of the bacteria are also becoming available worldwide. PCV15 is similar to PCV13 and protects against two additional types of the bacteria so may offer more protection.

This study, which lasts 2 months and is funded by Merck Sharp & Dohme (MSD), aims to assess if using PCV15 can protect against "carriage". To do this, investigators will use a well-established method already used with more than 2,000 people safely in other research. This involves "challenging" volunteers by putting a small amount of the pneumococcus bacteria into their noses. In this study, before they are challenged, volunteers will either be vaccinated with the real PCV15 vaccine or a dummy ("placebo"). The Investigators will then be able to compare the two groups to find out who the vaccine protected and who it did not.

After the study everyone who takes part and fit into certain criteria will be given antibiotics to clear the pneumococcus colonisation. They will also be regularly monitored during the study to ensure their safety.

A very small number of volunteers will be asked to have a biopsy to collect tissue samples from inside their nose before and after being vaccinated with PCV15. This will help researchers to understand more about how the immune system responds to the vaccine.

The information gain in this project will help the investigators to understand how exactly PCV15 vaccine protects people against pneumococcus. This means that this vaccine and future pneumococcal vaccines will be improved to protect many lives in future around the world.

DETAILED DESCRIPTION:
This is a Phase IV Double Blind (participant and observer) Placebo Controlled Randomised Controlled Trial (DBRCT) that will assess the superiority of PCV15 against placebo in healthy adults 18-50 years old exposed to an Experimental Human Pneumococcal Challenge (EHPC). Participants will be randomised 1:1 to receive PCV15 or placebo. We estimate a colonisation rate of 60% for the placebo group (84 participants with available endpoints, or up to 106 participants enrolled after adjusting for 20% attrition).

One month following randomisation and vaccination with PCV15 or placebo, all participants will be intranasally inoculated with Streptococcus pneumoniae serotype 3 (SPN3). Participants will be inoculated with a pure culture of a well-characterised, fully sequenced amoxicillin-sensitive pneumococcal serotype 3 (Clade Ia, strain LIV014-S3). Follow-up for 28 days will occur in the clinic with assessment of laboratory measures of the acquisition of nasal pneumococcal colonisation and of immune response after which participants will be required to take a 5-day course of antibiotics. Participants will be considered enrolled into the trial at vaccination.

Exploratory Nasal Biopsy cohort: From the 106 participants enrolled, 5 participants (not included in the primary endpoint sample size) will be asked to consent for a nasal biopsy procedure during screening visit and a second nasal biopsy 28 days after PCV15 vaccination. This cohort will not be blinded as only PCV15 will be provided. These participants wil not be inoculated and the study will terminate after the second biopsy visit (28 after vaccination).

The study is sponsored by the University of Oxford with two sites: Oxford (Centre for Clinical Vaccinology and Tropical Medicine) and Liverpool (Liverpool School of Tropical Medicine). The Experimental Human Pneumococcal Challenge model is well established on both sites.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 18 to 50 years old (inclusive) at the time of enrolment.
2. Medically healthy, such that according to investigator judgement, hospitalisation within the study period is not anticipated, and the participant appears likely to be able to remain a study participant through to the end of protocol-specified follow-up. Planned elective procedures for pre-existing conditions may be allowable.
3. Fluent spoken English - to ensure a comprehensive understanding of the research project and their proposed involvement.
4. Able to attend the scheduled visits and to comply with all study procedures, including internet access for the recording of electronic diary after inoculation.
5. Willing and able to give informed consent for participation in the study.
6. Willing to allow confirmation of past medical history either through provision of, or access to, a medical record summary or other medical documentation or allowing investigators to obtain a copy of their medical history from their GP practice or accessed via electronic patient records.
7. Willing to allow their GP and/or consultant, if appropriate, to be notified of participation in the study.
8. Willing to provide their national insurance number or passport number to be registered on The Over-Volunteering Prevention System (TOPS).
9. For participants of childbearing potential only: willing to use effective contraception for the duration of the study AND to have a pregnancy test on the day of screening and challenge.

Exclusion Criteria:

1. Research Participants:

   1. Participation in another research study, in which procedures performed could compromise the integrity of this study (such as significant volumes of blood taken), or are planning to do so within the trial period
   2. Currently a participant in a previous EHPC trial within the last 2 years or at the discretion of the study team
2. Vaccination (self-reported or confirmed from GP questionnaire or medical records/summary if deemed necessary at clinician discretion):

   1. Have had any previous pneumococcal vaccination in the past 5 years (including in a research study)
   2. Planned vaccination during the study
3. Allergy:

   1. Have an allergy to penicillin or amoxicillin (for main study cohort only)
   2. History of a bleeding disorder (e.g., Factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
   3. Have previous anaphylaxis or severe adverse reaction to any component/excipient of the vaccine or to any vaccine
   4. Allergy to Lidocaine local anaesthetic (for nasal biopsy cohort only)
4. Health History (self-reported or confirmed from GP questionnaire or medical records/summary if deemed necessary): moderate ill health including but not limited to:

   1. Asplenia or dysfuction of the spleen
   2. Chronic respiratory disease (e.g. asthma [on medication], COPD, emphysema, bronchiectasis)
   3. Chronic heart disease (e.g. angina, ischaemic heart disease, chronic heart failure) [controlled stable hypertension +/- angina may be included].
   4. Chronic kidney disease (e.g. nephrotic syndrome, kidney transplant, on dialysis)
   5. Chronic liver disease (e.g. cirrhosis, biliary atresia, hepatitis)
   6. Chronic neurological conditions
   7. Connective tissue disease
   8. Dementia
   9. Diabetes mellitus (including diet controlled)
   10. Immunosuppression or history of receiving immunosuppressive therapy - at the discretion of the investigator
   11. Individuals with cochlear implants
   12. Individuals with major cerebrospinal fluid leaks (e.g. following trauma, major skull surgery, or requiring CSF shunt)
   13. Recurrent otitis media.
   14. History of significant unexplained bleeding after a surgical or dental procedure (for nasal biopsy participants only)
   15. Have any uncontrolled medical/surgical/mental health conditions at the discretion of the study doctor.
   16. Major pneumococcal illness requiring hospitalisation within the last 10 years.
   17. Significant mental health condition (e.g previous admissions in a psychiatric unit, at the discretion of the clinician) that would impair the participant's ability to participate in the study
5. Taking Medications:

   1. Any medication that may affect the immune system in the last 3 months (e.g. systemic steroids [IM/IV], Roaccutane, disease modifying anti-rheumatoid drugs)
   2. Long-term use of antibiotics (see also section of Temporary Exclusion Criteria)
   3. Use of any medication or other product (prescription or over-the-counter) for symptoms of rhinitis or nasal congestion within the last 1 month
   4. Use of any medication affecting blood clotting (any oral/injectable anticoagulants)
6. Female participants who are pregnant, lactating or intending on becoming pregnant during the study
7. Direct caring role or close contact with individuals at higher risk of infection (for main study cohort only):

   1. Children under 5 years of age
   2. Chronic ill health or immunosuppressed adults
   3. Older adults
8. Smoker:

   1. Current or ex-smoker (regular cigarettes/cigars/e-cigarette/vaping/smoking of recreational drugs) in the last 6 months
   2. Previous significant smoking history (more than 20 cigarettes per day for 20 years or the equivalent [>20 pack years])
9. Suspected or known current alcohol or drug abuse, as per investigators discretion
10. Overseas travel during the follow-up period (from the time point of inoculation to antibiotic treatment or completion of the 28 day follow up period post inoculation)
11. Any other issue which, in the opinion of the study staff, may:

    1. Put the participant or their contacts at risk because of participation in the study
    2. Adversely affect the interpretation of the study results, or
    3. Impair the participant's ability to participate in the study
12. Study site staff or a partner or dependent child of study site staff

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of experimental SPN3 colonisation acquisition | Days 2, 7, 14 and 28 following experimental challenge
  Presence or absence of SPN3 bacteria detected by microbiological culture in nasal wash samples for 28 days after experimental SPN3 inoculation at 1-month post PCv15 vaccination compared with placebo.

SECONDARY OUTCOMES:
Density of experimental SPN3 colonisation | Days 2, 7, 14 and 28 following experimental challenge
  To determine the density CFU/ml of experimental SPN3 colonisation for 28 days following EHPC at 1-month post PCV15 vaccination by microbiological culture and molecular methods from nasal wash samples
Duration of experimental SPN3 colonisation | Days 2, 7, 14 and 28 following experimental challenge
  To determine the duration of experimental SPN3 colonisation for 28 days following EHPC at 1-month post PCV15 vaccination by classical culture and molecular methods from NW.
Vaccine-induced immune responses | Days 7 and 23 following vaccination and 2, 7, 14 and 28 following experimental challenge
  To compare vaccine-induced immune responses (antibody, antibody activity and B cells populations) to those who receive PCV15 versus control before and after experimental SPN3 challenge.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Drysdale, MRCPCH, PhD, PgDip PID, FRCPH, Principal Investigator — University of Oxford; Daniela M Ferreira, PhD, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Liverpool Vaccine Group, Liverpool, North West
  - Oxford Vaccine Group, Oxford, Oxfordshire

REFERENCES:
- [Derived] Macedo BR, Solorzano C, Hyder-Wright A, Lustosa Martinelli J, Robinson H, Brito-Mutunayagam S, Urban BC, Codreanu T, Elterish F, Mitsi E, Howard A, El Safadi D, Tanha K, Liu X, Mazur O, Ramasamy MN, Collins A, Ferreira DM, Drysdale SB. Protocol for a phase IV, Experimental Human Pneumococcal Challenge (EHPC) model to investigate Streptococcus pneumoniae serotype 3 (SPN3) colonisation following PCV15, a double-blind randomised controlled trial in healthy participants aged 18-50 years in the UK (RATIONALE-15). BMJ Open. 2025 Nov 24;15(11):e106028. doi: 10.1136/bmjopen-2025-106028. PMID 41290307